CLINICAL TRIAL: NCT01231282
Title: Technique Optimization and Anatomy of the Human Body With Whole-body Diffusion-weighted MRI: Study With Healthy Volunteers
Brief Title: Technique Optimization With Whole-body Diffusion-weighted MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: S52777
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2010-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diffusion-weighted MRI (Experimental): MRI
  Interventions: Other: diffusion-weighted MRI

INTERVENTIONS:
Other: diffusion-weighted MRI — MRI scan without contrast administration and without radiation exposure

SUMMARY:
Whole body diffusion-weighted imaging is a functional magnetic resonance imaging technique that characterizes tissue by probing changes in water diffusion secondary to differences in the tissue microstructure. These changes in water diffusion result in differences in signal intensity on diffusion-weighted images that are quantified with the apparent diffusion coefficient (ADC). In malignant lesions, the extravascular extracellular space (EES) will be diminished, due to the increased number of cells. This will restrict water diffusion, identified by increased signal intensity (SI) on native diffusion-weighted images and low ADC. Contrary, in tissue with low cellularity, like benign lesions and treatment induced necrosis, the EES will be enlarged due to the lower density of cells, or in case of necrosis, the complete absence of cellular organization. This will facilitate water diffusion, leading to absent SI on native diffusion-weighted images and high ADC.

The purpose of this study is to image anatomy and lymph nodes in healthy volunteers with whole body diffusion-weighted imaging. This way maps of normal anatomy can be created on the whole body diffusion-weighted images which can be used as a reference in further studies with patients scanned with the same whole body diffusion-weighted imaging scan protocol.

A group of 30 healthy volunteers will receive a whole body diffusion-weighted imaging scan on a 3 Tesla T-MRI system.

A total scan session will take about 30 minutes. Contrast administration is not required and patients will not be exposed to radiation.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* no severe illness in the past
* no current infection/inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
normal aspect of human anatomy on WB-DWI images/ technique optimization | up to 12 months
  assessment after all the scans of the healthy volunteers are collected

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Vandecaveye, Principal Investigator — vincent.vandecaveye@uzleuven.be
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] De Paepe KN, Van Keerberghen CA, Agazzi GM, De Keyzer F, Gheysens O, Bechter O, Wolter P, Dierickx D, Janssens A, Verhoef G, Oyen R, Koole M, Vandecaveye V. Quantitative Whole-Body Diffusion-weighted MRI after One Treatment Cycle for Aggressive Non-Hodgkin Lymphoma Is an Independent Prognostic Factor of Outcome. Radiol Imaging Cancer. 2021 Mar 26;3(2):e200061. doi: 10.1148/rycan.2021200061. eCollection 2021 Mar. PMID 33817648